CLINICAL TRIAL: NCT04380376
Title: Single-center, Prospective, Open-label, Comparator Study, Blind for Central Accessor to Access the Efficacy, Safety, and Tolerability of Inhalations of Low-doses of Melphalan in Patients With Pneumonia With Confirmed or Suspected COVID-19
Brief Title: Low-doses Melphalan Inhalation in Patients With COVID-19 (CoronavIrus Disease 2019) Pneumonia
Acronym: MICOV
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal State Budgetary Institution, Pulmonology Scientific Research Institute (Other Government)
Collaborators: Medsi Clinic #1, Moscow (Other); Moscow State University of Medicine and Dentistry (Other)
Responsible Party: Principal Investigator, Kirill Zykov, Deputy director for Science and Innovations, Federal State Budgetary Institution, Pulmonology Scientific Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSRI05-20
Record Dates: First submitted 2020-05-06; First posted 2020-05-08 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; Viral Pneumonia
Keywords: COVID; treatment; inhalation; alkylating drug; pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia, Viral; Respiratory Aspiration; Pneumonia | interventions — Melphalan; Standard of Care

STUDY DESIGN:
Intervention Model Description: Prospective, Single-center, Open-Label, Central Assessor Blinded, Comparative Study
Who Masked: Outcomes Assessor
Masking Description: An independent central blinded assessor will be blinded to study treatment and will review the clinical response assessments. In case of a discrepancy with the Investigator's assignment of clinical response, the adjudication committee's assessment will prevail.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melphalan inhalations (Experimental): Inhalations with Melphalan 0,1 mg dissolved in 2 ml sodium chloride (NaCl) 0,9% 1 per day for 7-10 consequent days
  Interventions: Drug: Melphalan
- Standard of care group (Other): Patients assigned to the standard of care group will not receive any additional therapy.
  Interventions: Other: Standard of care

INTERVENTIONS:
Drug: Melphalan — Inhalations with low doses of Melphalan for 7-10 consequent days
  Other Names: Alkeran
  Arms: Melphalan inhalations
Other: Standard of care — the patients will receive only SOC (standard of care) treatment
  Arms: Standard of care group

SUMMARY:
This single-center, prospective, open-label, comparator study, blind for central accessor evaluates the efficacy, safety of inhalations of low-doses of melphalan in patients with pneumonia with confirmed or suspected COVID-19. All patients will receive 0,1 mg of melphalan in 7-10 daily inhalations 1 time per day.

DETAILED DESCRIPTION:
It was previously shown that in ultra-low (more than 100 times lower than conventional therapeutic) doses inhalations of alkylating drug (melphalan) are effective in severe steroid-resistant bronchial asthma, a form of the disease often characterised by neutrophilic type of inflammation. The exacerbation frequency reduced after the treatment, steroid-sparing effect was shown, morphological signs of bronchial epithelial regeneration were revealed and quality of life of asthmatic patients, treated with ultra-low doses of melphalan, improved. In preclinical studies and studies with volunteers, it was found that inhalations of ultra-low doses of melphalan do not have cytotoxic properties, but have local and systemic anti-inflammatory effects and decrease the activation of lymphocytes due to blockade of heavy β-chain of the interleukin (IL)-2 surface receptor. In addition, in ultra-low concentrations, alkylating agents are able to disrupt the cell signalling through the receptor for tumor necrosis factor (TNF), thereby exerting a protective effect from the cytotoxic activity of TNF-α, which leads to the anti-inflammatory response.

Taking into account, that severe cases of COVID are characterised with hyperergic inflammatory response (and in some cases even with the development of "cytokine storm") it can be assumed that the inhalation use of low-doses of melphalan due to its anti-inflammatory properties can be effective treatment for patients with COVID-associated pneumonia.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. A patient must have confirmed the diagnosis of bi-lateral moderate / severe pneumonia ( viral or viral-bacterial with confirmed of suspected COVID-19).
3. Presence new infiltrates or increase already available infiltrates of pulmonary infiltrates on lung CT within 48 hours before baseline.
4. A patient has as minimum one of the following symptoms:

fever >38 degrees Celsius, cough, dyspnea, SaO2 (arterial oxygen saturation) <95% (with room air)

Exclusion Criteria:

1. Informed consent is withdrawn by the patient.
2. The patient doesn't follow the instructions of the research staff regarding the requirements of the research protocol.
3. Unable to contact the patient.
4. The researcher believes that participation in the study is not in the interests of the patient and / or further participation in the study is unsafe for the patient's health.
5. There is a violation of the criteria for inclusion and / or non-inclusion in the study.
6. The patient has developed an adverse event, which, according to the researcher, makes further participation in the study unsafe for the patient.
7. The licensing authority or ethics committee, for any reason, decides to discontinue the entire study or close this research center.
8. A female patient becomes pregnant, is planning a pregnancy, or is breastfeeding while participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
The changes of COVID Ordinal Outcomes Scale | baseline vs Day 14, day 28
  The number of patients with the clinical improvement is defined as an improvement of two points (from the status at baseline) on an ordinal scale of clinical improvement on day 28 or discharge from hospital ( whatever occurs earlier)
  1. Death
  2. Hospitalized with Invasive mechanical ventilation plus additional organ support - ECMO / pressors / RRT
  3. Hospitalized with intubation and mechanical ventilation
  4. Hospitalized on non-invasive ventilation or high flow oxygen.
  5. Hospitalized on a mask or nasal prongs.
  6. Hospitalized no oxygen therapy.
  7. Ambulatory, with limitation of activities.
  8. Ambulatory, no limitation of activities. I. No clinical or virological evidence of infection.
Percentage of the patients with Clinical Recovery | baseline vs day 7, day 14, day 28
  Percentage of the patients with clinical recovery which is defined as a normalisation of fever, respiratory rate, and oxygen saturation, and improvement of cough, sustained for at least 72 hours, or live hospital discharge, whichever comes first.
  Normalization and improvement criteria:
  * Fever - <37°C,
  * Respiratory rate - ≤24/minute on room air,
  * Oxygen saturation - >94% on room air,
  * Cough - mild or absent on a patient reported scale of severe, moderate, mild, absent.
The changes of the Borg's scale | Baseline vs day 7, day 14, day 28
  The evaluation of changes in modified Borg dyspnea scale. From 0 to 10 units.A lower score means a better clinical result (0 is the absence of dyspnea, and 10 - is maximal dyspnea). Minimal clinically important difference is 1 unit.

SECONDARY OUTCOMES:
CRP level | baseline, day 7, Day 14, Day 28
  Change in C-reactive protein (CRP) level from baseline in mg/ml. A lower level of CRP means a better clinical result.
Lymphocyte count | baseline, day 7, Day 14, Day 28
  Change in blood absolute lymphocyte count from baseline. A higher number of lymphocytes means a better clinical result.
D-dimer | baseline, day 7, Day 14, Day 28
  Change in blood D-dimer level from baseline. A lower level of D-dimer means a better clinical result.
IL-6 | baseline, day 7, Day 14, Day 28
  Change in peripheral blood IL-6 level from baseline. A lower level of IL-6 means a better clinical result.
Percentage of patients without artificial lung ventilation | baseline, day 7, Day 14, Day 28
  Percentage of patients without artificial lung ventilation during the study. A lower percentage of patients means a better clinical result.

CONTACTS AND LOCATIONS:
Overall Officials: Kirill A Zykov, Prof, Principal Investigator — Federal State Budgetary Institution, Pulmonology Scientific Research Institute
Locations (2):
- Russia (2):
  - Kirill Zykov, Moscow
  - Clinical hospital, Moscow

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pukhalsky AL, Shmarina GV. Stimulatory and protective effects of alkylating agents applied in ultra-low concentrations. Pharmacology. 2001;62(3):129-32. doi: 10.1159/000056084. PMID 11287812
- [Background] Pukhal'skii AL, Shmarina GV, Zykov KA, Aleshkin VA. [Effect of steroid therapy on the clinical course of bronchial asthma]. Vestn Ross Akad Med Nauk. 2009;(6):3-9. Russian. PMID 19645099
- [Background] Pukhalsky A, Shmarina G, Alioshkin V, Sabelnikov A. Alkylating drugs applied in non-cytotoxic doses as a novel compounds targeting inflammatory signal pathway. Biochem Pharmacol. 2006 Nov 30;72(11):1432-8. doi: 10.1016/j.bcp.2006.03.008. Epub 2006 Mar 14. PMID 16620792